CLINICAL TRIAL: NCT01426789
Title: A Multicenter, 12 Week, Randomized, Double-blind, Placebo-controlled Biomarker Study of Secukinumab (AIN457) in Rheumatoid Arthritis Patients Followed by an Open Label Extension
Brief Title: A Biomarker Study of Secukinumab in Rheumatoid Arthritis (RA) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457F2208
Record Dates: First submitted 2011-08-12; First posted 2011-08-31 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; IgG1K monoclonal antibody; Interleukin-17A neutralizing
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Secukinumab (Experimental): 10 mg/kg intravenous (I.V.)
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo I.V.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo to secukinumab I.V.
  Arms: Placebo
Drug: Secukinumab — In part 1 (blinded period), participants randomized to secukinumab received 10 mg/kg I.V.. Participants, enrolled in part 2 (open label), received secukinumab 300 mg subcutaneous.
  Other Names: AIN457
  Arms: Secukinumab

SUMMARY:
This study aims to confirm if patients with a specific biomarker might have a better response to secukinumab treatment. To meet this purpose, exploratory biomarker studies will be done. The goals of these exploratory studies are to (1) find biomarkers that will identify persons with rheumatoid arthritis who will have the best possible response to secukinumab and (2) to identify persons who will have fewer side effects in order to maximize their benefit from secukinumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis
* Patients must be either DMARD naive or have failed at least one DMARD agent (e.g. MTX, leflunamide or sulfasalazine)
* Patients are allowed up to 3 DMARDs at study entry (e.g. MTX, sulfasalazine or hydroxychloroquine) as long as their dose was stable for 4 weeks prior to initiating study treatment
* Disease activity at screening defined by ≥6 out of 28 tender joints and ≥6 out of 28 swollen joints and hsCRP >10mg/L

Exclusion Criteria:

* Patients with severe rheumatoid arthritis (functional status class IV according to the ACR 1991 revised criteria)
* Previous exposure to secukinumab or any other biologic, including TNF inhibitors.
* Use of high potency opioid analgesics
* Pregnant or nursing (lactating) women
* Use of any investigational drug other than RA therapy and/or devices at the time of randomization or within 30 days or 5 half-lives of randomization, whichever is longer.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- United States (16):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tuscon, Arizona
  - Novartis Investigative Site, Anahiem, California
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Coral Gables, Florida
  - Novartis Investigative Site, Fleming Island, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pinellas Park, Florida
  - Novartis Investigative Site, Venice, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, South Bend, Indiana
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Statesville, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, San Antonio, Texas
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Kortrijk
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
- Russia (7):
  - Novartis Investigative Site, Smolensk, Russia
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Yaroslavl
- United Kingdom (2):
  - Novartis Investigative Site, Manchester, Manchester
  - Novartis Investigative Site, Belfast

REFERENCES:
- [Derived] Burmester GR, Durez P, Shestakova G, Genovese MC, Schulze-Koops H, Li Y, Wang YA, Lewitzky S, Koroleva I, Berneis AA, Lee DM, Hueber W. Association of HLA-DRB1 alleles with clinical responses to the anti-interleukin-17A monoclonal antibody secukinumab in active rheumatoid arthritis. Rheumatology (Oxford). 2016 Jan;55(1):49-55. doi: 10.1093/rheumatology/kev258. Epub 2015 Aug 12. PMID 26268815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a 12 week, randomized, double blind phase (part 1), a 40 week, open label phase (part 2), and a 3 month safety follow-up. Participants from the secukinumab arm, who completed part 1 and had an ACR50 or greater response at week 12, and participants from the placebo arm, who completed part 1, were eligible for the open label phase.
Pre-assignment Details: One hundred participants received study treatment in part 1. Ten participants discontinued during part 1. At the end of part 1, 76 participants were eligible to take secukinumab treatment in part 2.
Groups:
- Group 1: Part 1: secukinumab 6 x 10 mg/kg i.v.; Part 2: secukinumab 300 mg sc monthly
- Group 2: Part 1: secukinumab 6 x 10 mg/kg i.v.; part 2: no study treatment
- Group 3: Part 1: placebo; Part 2: secukinumab 4 x 300 mg sc loading dose (at weeks 12, 13, 14 and 16), then 300 mg sc monthly
- Group 4: Part 1: placebo; Part 2: no study treatment
Period: Part 1
Arm/Group | Secukinumab | Placebo | Group 1 | Group 2 | Group 3 | Group 4
Started | 68 | 32 | 0 | 0 | 0 | 0
Completed | 62 | 28 | 0 | 0 | 0 | 0
Not Completed | 6 | 4 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Secukinumab | Placebo | Group 1 | Group 2 | Group 3 | Group 4
Started | 0 | 0 | 49 | 13 | 27 | 1
Completed | 0 | 0 | 34 | 12 | 19 | 1
Not Completed | 0 | 0 | 15 | 1 | 8 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Administrative problems | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 5 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 68 | 32 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (11.45) | 54.5 (10.30) | 51.1 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 25 | 73
  Male | 20 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve American College of Rheumatology Response of 20 (ACR20 ) in Association With the Presence or Absence of the HLA-DRB1 *4 Allelic Group
Description: A participant was considered to be a responder according to the ACR20 criteria if the participant had at least 20% improvement in both the tender joint count and swollen joint count measures, and in at least 3 of the following 5 measures: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score, and/or C-reactive protein (CRP)/Erythrocyte Sedimentation Rate (ESR).
Time Frame: 12 weeks
Population: Participants, who completed part 1, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 62 | 28
Percentage of participants
  HLADRB1 *04 carriers | 45.2 | 10.7
  HLADRB1 *04 non-carriers | 41.9 | 14.3

2. Primary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) in Association With the Presence or Absence of HLA-DRB1 04
Description: The DAS28 is a measure of disease activity in RA. The score is calculated by a complex mathematical formula, which includes the tender joint count(TJC) and swollen joint count (SJC) out of a total of 28 joints, the high-sensitivity C-reactive protein (hsCRP), and the subject's 'global assessment' of disease activity/general health (GH). The subject's global assessment/GH was indicated by a visual analogue scale of 100 mm where the participant marked a point on a 100 mm line between 0 and 100 (0 indicated very good and 100 indicated very bad). The following formula was used to calculate DAS28: DAS-CRP = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) = 0.36*ln(CRP+1) + 0.014*GH = 0.96. A DAS28-CRP score > 5.1 implies active disease, <3.2 implies controlled disease and <2.6 implied remission. A negative change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Participants, who completed part 1, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 62 | 28
score on a scale
  HLA-DRB1 *04 carriers | -2.5 (0.5273) | -0.6 (0.5750)
  HLA-DRB1 *04 non-carriers | -2.2 (0.5618) | -0.8 (0.6098)

3. Secondary Outcome: Percentage of Participants Who Achieve ACR50 and ACR70 With the Presence/Absence of the HLA-DRB1*04 Allelic Group
Description: A participant was considered to be a responder according to the ACR50 or ACR70 criteria if the participant had at least 50% or 70% improvement, respectively, in both the tender joint count and swollen joint count measures, and in at least 3 of the following 5 measures: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score, and/or C-reactive protein (CRP)/Erythrocyte Sedimentation Rate (ESR).
Time Frame: 12 weeks
Population: Participants, who completed part 1, were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 62 | 28
Percentage of participants
  ACR50: HLADRB1 *04 presence | 38.7 | 7.1
  ACR50: HLADRB1 *04 absence | 35.5 | 10.7
  ACR70: HLADRB1 *04 presence | 8.1 | 0.0
  ACR70: HLADRB1 *04 absence | 8.1 | 7.1

4. Secondary Outcome: Change From Baseline in DAS28 in Association With the Presence or Absence of HLA-DRB1 *SE (Positive), HLA-DRB1 *401 (Carrier) and HLA-DRB1 Position 11 V/L and in Association With Other Biomarkers
Description: as for outcome 2
Time Frame: baseline, 12 weeks
Population: Participants, who completed part 1, were included in the analysis. Statistical analysis was not done on the other biomarkers: osteoprotegerin (OPG), rheumatoid factor (RF), anti-cyclic citrullinated peptide antibodies (CCP) and hsCRP. Therefore, data is provided for the alleles only.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 62 | 28
score on a scale
  HLA-DRB1 *SE carrier | -2.6 (0.5049) | -0.5 (05240)
  HLA-DRB1 *SE non-carrier | -2.3 (0.5376) | -2.2 (0.6977)
  HLA-DRB1 *0401 carrier | -2.4 (0.5922) | 0.1 (0.7503)
  HLA-DRB1 *401 non-carrier | -2.3 (0.5133) | -0.9 (0.5456)
  HLA-DRB1 position 11 V/L carrier | -2.5 (0.4901) | -0.4 (0.5218)
  HLA-DRB1 position 11 V/L non-carrier | -2.2 (0.5706) | -2.2 (0.6954)

ADVERSE EVENTS:
Description: Adverse events that occurred in subjects after they discontinued during or at the end of Part 1 are not included in the Part 2 safety analysis. Therefore, treatment groups from Part 1 and groups 1 and 3 from Part 2 are presented only.
Groups:
- Secukinumab: 10mg/kg i.v.
Arm/Group | Secukinumab | Placebo | Group 1 | Group 3
Serious Adverse Events (participants affected / at risk) | 4/68 | 2/32 | 4/49 | 4/27
Other Adverse Events (participants affected / at risk) | 13/68 | 9/32 | 15/49 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=68) | Placebo (N=32) | Group 1 (N=49) | Group 3 (N=27)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Vasculitis necrotising (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=68) | Placebo (N=32) | Group 1 (N=49) | Group 3 (N=27)
Dry eye (Eye disorders) | 1 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Blood pressure increased (Investigations) | 0 | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.